CLINICAL TRIAL: NCT05827146
Title: Double-blinded, Placebo-controlled, Munticenter, Phase IIa Clinical Trial of Hepalatide in Patients With Chronic Hepatitis D
Brief Title: Study of Hepalatide in Chronic Hepatitis D(CHD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L47-HD-IIa
Record Dates: First submitted 2023-02-17; First posted 2023-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Chronic Hepatitis D Infection
Keywords: chronic hepatitis D; hepalatide; hepatitis D virus
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hepalatide 2.1mg (Experimental): 2.1 mg/day subcutaneously (s.c.) for 4 week
  Interventions: Drug: Hepalatide
- Hepalatide 4.2mg (Experimental): 4.2 mg/day subcutaneously (s.c.) for 4 week
  Interventions: Drug: Hepalatide
- Hepalatide 6.3mg (Experimental): 6.3 mg/day subcutaneously (s.c.) for 4 week
  Interventions: Drug: Hepalatide
- Placebo 2.1mg/4.2mg/6.3mg (Placebo Comparator): Placebo 2.1 mg/4.2mg/6.3mg, once a day subcutaneously (s.c.) for 4 week
  Interventions: Drug: Hepalatide Placebo

INTERVENTIONS:
Drug: Hepalatide — Either the placebo or hepalatide (2.1 mg, 4.2 mg, or 6.3 mg) will be given for 4 consecutive weeks. s.c., once daily.
  Other Names: L47
  Arms: Hepalatide 2.1mg; Hepalatide 4.2mg; Hepalatide 6.3mg
Drug: Hepalatide Placebo — Either the placebo or hepalatide (2.1 mg, 4.2 mg, or 6.3 mg) will be given for 4 consecutive weeks. s.c., once daily.
  Other Names: Placebo
  Arms: Placebo 2.1mg/4.2mg/6.3mg

SUMMARY:
A phase 2a clinical Study of Hepalatide for Injection in Subjects with Chronic Hepatitis D

DETAILED DESCRIPTION:
This is a four-arm parallel-group, randomized, placebo-controlled, double-blind, multicenter Phase IIa clinical trial. The CHD subjects who meet the eligibility criteria will be randomly assigned 1:1:1:1 to receive either the placebo or investigational drug (2.1 mg, 4.2 mg, or 6.3 mg), with 6 subjects per group . The placebo or the corresponding dose of the investigational drug will be given for 4 consecutive weeks, followed by a 4-week follow-up period. Subjects will be given entecavir for the treatment of hepatitis B infection during and after the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years old (both inclusive);
* HBsAg (+) and/or HBV DNA (+) for at least 6 months (clinically diagnosed as "chronic hepatitis B");
* HDV-antibody (IgG/IgM) (+) and HDV RNA (+);
* 1×ULN <ALT<10×ULN；
* Patients with hepatitis B eligible to receive treatment with NAs according to current guidelines for the diagnosis and treatment of hepatitis B;
* Patients who do not plan a pregnancy within two years (women who are not pregnant or lactating) and agree to take effective contraceptive measures throughout the treatment period and within 3 months after the last dose;
* Patients who did not participate in any other clinical trials within 3 months;
* Patients with good compliance with the study protocol;
* Patients who understand and agree to sign an informed consent form.

Exclusion Criteria:

* Decompensated liver disease: Direct bilirubin > 1.2× ULN, prothrombin time > 1.2× ULN, and serum albumin < 35 g/L;
* Patients with abnormal results of routine hematology test: White blood cell count (WBC) < 3×109/L, neutrophil count < 1.5×109/L and platelet count < 60×109/L;
* Severely decompensated hepatic fiborosis or decompensated cirrhosis: Definitely diagnosed decompensated cirrhosis by imaging examinations such as a Color Doppler ultrasound and CT of the abdomen or clinically diagnosed decompensated cirrhosis by the investigator, or a Metavir fibrosis score of 4 on a liver biopsy sample, or a Child-Pugh score > 7 for liver function assessment;
* Patients who have any of the following conditions:

  1. A history of decompensated liver disease (ascites, jaundice, hepatic encephalopathy, variceal bleeding);
  2. A history of serious cardiovascular disease (including unstable or uncontrolled cardiovascular disease within 6 months);
  3. Serious mental illness or a history of serious mental illness;
  4. A history of organ transplantation;
  5. Uncontrolled epilepsy, mental illness, or poorly controlled diabetes or hypertension;
  6. Autoimmune disease, immune-related extrahepatic manifestations (vasculitis, purpura, arteritis nodosa, peripheral neuropathy, and glomerulonephritis), thyroid disease, malignant tumor, and receiving immunosuppressive therapy;
  7. Underlying diseases such as severe infection, heart failure, chronic obstructive pulmonary disease, and other severe diseases;
  8. A history of alcohol or drug abuse.
* Creatinine clearance < 60 mL/min;
* HAV/HCV/HEV/HIV co-infection;
* Resistance to or poor response to Entecavir;
* An allergic reaction to Entecavir;
* Patients who have used interferon within 3 months before the screening period;
* Previously received L47 or Bulevirtide;
* Women who have a positive pregnancy test;
* Patients who have other significantly abnormal results of laboratory or auxiliary tests and are unsuitable for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Hepatitis D Virus(HDV) RNA level | Week 4
  HDV RNA level at week4

SECONDARY OUTCOMES:
Change in Alanine transaminase(ALT) from baseline | Week 4
  Changes in ALT values at Week 4 compared to baseline
Change in HDV RNA from baseline | Week 4
  Changes in HDV RNA levels at Week 4 compared to baseline

OTHER OUTCOMES:
ALT level | Week 4
  ALT level at Week 4
Number of Participants With ALT normalization | Week 4
  Number of Participants With Normal ALT at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University
Locations (3):
- China (2):
  - The first affiliated hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The first hospital of Jilin University, Changchun
- the National cancer center of Mongolia, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No